CLINICAL TRIAL: NCT03985020
Title: Super HEROES: Searching How the Extract Rebaudioside Occludes Excess Steatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Tania Mitsinikos, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-19-00212
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three possible groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): The control group will receive standard of care dietary advice for their solid food and beverage intake.
- Water Intervention (Active Comparator): We will order and deliver bottled water to the homes of subjects in the treatment group. We will provide each participant with a weekly supply of about 36 16.9 fl oz single-serving containers. We will instruct subjects to notify us by calling a dedicated telephone line on occasions when a delivery is expected but not received so that the problem can be corrected expeditiously.
  Interventions: Other: Water Intervention
- Stevia Intervention (Experimental): We will order and deliver a commercially-available stevia-sweetened soft drink Zevia (Los Angeles, CA) to each participant in the treatment group. We will provide each participant with a weekly supply of 24 12 fl oz single-serving containers. Zevia will be provided in an assortment of flavors for the first week, then catered to the preference of the participant for the remainder of the study. We will instruct subjects to notify us by calling a dedicated telephone line on occasions when a delivery is expected but not received so that the problem can be corrected expeditiously. Participants will also be asked to keep track of how many containers they consume using a sticker chart, and we will also phone parents weekly to verify the sticker charts
  Interventions: Other: Stevia Intervention

INTERVENTIONS:
Other: Stevia Intervention — We will use commercially available stevia sweetened soft drink Zevia.
  Arms: Stevia Intervention
Other: Water Intervention — Bottled Water
  Arms: Water Intervention

SUMMARY:
In order to determine whether rebaudioside consumption can be used as a treatment for adolescents with Non-alcoholic Fatty Liver Disease (NAFLD) by demonstrating a decrease in alanine aminotransferase (ALT) levels participants will be randomized to receive one of three 8-week liquid diet interventions:

1. Standard of care
2. Water delivery
3. Water with Rebaudioside (stevia natural sweetener)

DETAILED DESCRIPTION:
Rationale: Current treatment strategies for Nonalcoholic fatty liver disease, NAFLD, have focused on lifestyle management through a combination of diet and exercise but there are no recommendations for dietary changes that have been proven superior to others. Preliminary data showing an improvement in liver enzymes and fibrosis in mice has demonstrated a novel use of rebaudioside, the non-caloric sweetener (NCS) Stevia leaf's extract, potentially identifying this NCS as a therapeutic intervention where currently there are no targeted treatments.

Intervention: All participants will receive standard of care for diet and nutrition. Additionally, participants will be randomized to one of four 8-week liquid diet interventions:

1. Standard of Care
2. Water Delivery
3. Water with Rebaudioside (Stevia Natural Sweetener)

Objectives and Purpose: To determine whether rebaudioside consumption can be used as a treatment for adolescents with NAFLD by demonstrating a decrease in ALT levels.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-18 years
* ALT > 45 IU/L (twice the normal amount)
* BMI >85%
* Fat >5% and kPa> 2.7

Exclusion Criteria:

* Physician diagnosis of a major medical illness including, but not limited to, chronic liver disease, immunodeficiency disorder, hypothalamic obesity, or a genetic cause of obesity.
* Familial hyperlipidemia
* Positive hepatitis lab
* Antibiotics within 1 month of beginning the study
* Physical, mental, or cognitive issues preventing participation
* Pregnancy
* Smoking or drinking

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Alanine Transaminase (ALT) | Week 1 to week 8 (IU/L)
  A fasting blood sample will be taken at baseline and week 8 and assess change over time in all 3 groups

SECONDARY OUTCOMES:
Change in Fat percentage | week 1 to 8 weeks (%)
  Measured using DEXA
Change in kPA levels | week 1 to 8 weeks (kPA)
  Measured using MR elastography (non-sedated study)
Change in Height | week 1 to 8 weeks (cm)
  Height will be measured in duplicate within .5cm.
Change in Weight | week 1 to 8 weeks (kg)
  Measured using an electric scale.
Change in Waist Circumference | week 1 to 8 weeks (cm)
  Hip-to-waist ratio will be calculated using a measuring tape that does not stretch, measuring twice at hip-level and twice at waist-level and averaging the results
Change in Acanthosis nigricans skin exam | week 1 to 8 weeks
  An Acanthosis Nigricans (AN) skin exam will be performed at each visit. Acanthosis Nigricans is an indicator for disorders of insulin resistance.
Change in Triglyceride levels | week 1 to 8 weeks
  measured by fasting blood sample
Change in Glucose Level | Week 1 to week 8 (mg/dl)
  Measured by fasting blood samples
Change in Insulin Level | Week 1 to week 8 (UIU/mL)
  Measured by fasting blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Tania Mitsinikos, MD, Principal Investigator — Children's Hospital Los Angeles; Rohit Kohli, MBBS, MS, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States